CLINICAL TRIAL: NCT02101723
Title: Effects of Sprinkles With and Without Iron on Zinc Absorption From Local Foods in Kenyan Toddlers, Including the Gut Microbiome
Brief Title: Effect of Sprinkles With and w/o Fe on Zn Absorption in Kenyan Toddlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); International Atomic Energy Agency (Other Government); Moi University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 11-0227; K24DK083772 (NIH); 15827 (Other Grant/Funding Number: IAEA); 16933 (Other Grant/Funding Number: IAEA)
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Micronutrient Deficiencies
Keywords: Zinc absorption; Micronutrient supplement; Microbiome; Kenya; Complementary foods; Home fortification

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Micronutrient Powder (MNP) + Zn/Fe (Active Comparator): Micronutrient Powder with 5 mg Zn and 12 mg Fe
  Interventions: Dietary Supplement: MNP + Zn/Fe
- MNP + Zn (Active Comparator): Micronutrient Powder with 5 mg Zn
  Interventions: Dietary Supplement: MNP + Zn
- Control (Placebo Comparator): Placebo sachets without micronutrients
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: MNP + Zn/Fe — Micronutrient powder with 12 mg Fe and 5 mg Zn provided daily from 6-9 months of age
  Arms: Micronutrient Powder (MNP) + Zn/Fe
Dietary Supplement: MNP + Zn — Micronutrient powder with 5 mg Zn provided daily from 6-9 months of age
  Arms: MNP + Zn
Dietary Supplement: Placebo — Placebo powder without micronutrients
  Arms: Control

SUMMARY:
The investigators propose to study the effects of increased iron intake by home fortification of complementary foods on the gastrointestinal microbial development, inflammatory responses, and zinc (Zn) absorption. The proposed subjects are 9 month olds living in a malaria endemic area of rural Kenya who are randomized at 6 months of age to one of three fortificant groups: 1) Sprinkles™ with 12mg Iron(Fe)/day + other micronutrients, including 5mg/d Zn (test); Sprinkles™ with 0 mg/d Fe + other micronutrients, including 5mg/d Zn (control); Sprinkles™ with no micronutrients (placebo). The investigators hypothesize that the microbiome will be significantly different in the three groups and that Zn absorption and status, in addition to immune and oxidant status will be improved in the non-Fe fortified groups when compared to the Fe-fortified group.

DETAILED DESCRIPTION:
Specific aims include exploration of possible mechanisms of adverse events that have been observed in iron supplementation trials in infants in malaria endemic regions by:

1. Characterizing the impact of enteral iron administration on the evolution of the intestinal microbiome in infants from 6 to 9 months of age.
2. Characterizing iron administration-associated inflammatory responses and correlate these with changes in the intestinal microbiome in infants from 6 to 9 months of age. Specifically, changes in the microbiome will be correlated with biomarkers reflecting:

   1. Intestinal inflammation;
   2. Systemic inflammation, bacterial translocation, and oxidant stress;
   3. Iron status and homeostasis
3. Quantify to what degree Fe interferes with Zn absorption (TAZ) and how it affects the size of the infant's exchangeable zinc pool (EZP).

ELIGIBILITY:
Inclusion Criteria:

* Term infant
* Birthweight > 2500 g
* Healthy with no apparent congenital anomalies
* Up-to-date with vaccinations
* Hb >10 g/dL
* Breastfeeding with intent to continue for duration of study
* Negative blood slide for malaria
* Written informed consent

Exclusion Criteria:

* Acute malnutrition
* Current or anticipated used of infant formula or other fortified products
* Current or planned use of iron (or zinc) supplements
* Previous hospitalization for malaria within the last four weeks
* Persistent diarrhea

Ages: 5 Months to 10 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Changes in GI microbiome | 6 and 9 months of age
  Identify and quantify the phylogenic distribution of bacterial genera in the infants from 6 to 9 months in prevalence or abundance with iron supplementation at baseline, mid-point and 9 months.

SECONDARY OUTCOMES:
Change in Biomarkers of intestinal and system inflammation | 6 and 9 months of age
  Compare mean baseline and 9 month values biomarkers of intestinal and systemic inflammation and look at differences among the 3 groups.
Absorption of Zn | 9 months of age
  Determine the effects of increased iron intake on zinc absorption from micronutrient powder added to local complementary foods of Kenyan toddlers in a malaria-endemic area.
Size of exchangeable Zn pool | 9 months of age
  Determine the effect of increase iron intake on size of exchangeable Zn pool (EZP) after 3 months of home fortification with micronutrient powder in maize-based diets in rural Kenyan infants.
Change in Biomarkers of bacterial translocation | 6 and 9 mo of age
  To compare biomarkers of bacterial translocation among the 3 groups and look at longitudinal differences between 6 and 9 mo of age.
Change in Biomarkers of oxidative stress | 6 and 9 mo of age
  Compare biomarkers of oxidative stress among the 3 groups and look at longitudinal differences at 6 and 9 mo of age.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy F Krebs, MD, Principal Investigator — University of Colorado, Denver; Fabian Esamai, MD, Study Director — Moi Univeristy
Locations (2):
- University of Colorado Denver, Aurora, Colorado, United States
- Moi University, Eldoret, Kenya

REFERENCES:
- [Background] Esamai F, Liechty E, Ikemeri J, Westcott J, Kemp J, Culbertson D, Miller LV, Hambidge KM, Krebs NF. Zinc absorption from micronutrient powder is low but is not affected by iron in Kenyan infants. Nutrients. 2014 Dec;6(12):5636-51. doi: 10.3390/nu6125636. PMID 25493942